CLINICAL TRIAL: NCT00646412
Title: A Prospective, Randomised, Controlled, Single-blind Phase I-II Clinical Trial on the Safety of A-Part® Gel as Adhesion Prophylaxis After Major Abdominal Surgery Versus a Non-treated Group
Brief Title: A-Part® Gel as Adhesion Prophylaxis After Major Abdominal Surgery Versus a Non-treated Group
Acronym: A-PART
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAG-G-H-0602
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Adhesions; Abdominal Cavity
Keywords: randomized, controlled, single-blind study; Adhesion Prophylaxis; Abdominal Surgery; Laparotomy, median
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): A-Part® Gel
  Interventions: Device: A-Part® Gel
- B (No Intervention): untreated control group

INTERVENTIONS:
Device: A-Part® Gel — 10 - 20 ml of A-Part® Gel will be administered before abdominal wall closure in a standardised fashion
  Arms: A

SUMMARY:
The safety of applying A-Part® Gel intra-peritoneally under the incision in order to prevent post-surgical adhesions after median laparotomy.

DETAILED DESCRIPTION:
Primary Objective:

• first assessment of the safety of applying A-Part® Gel as adhesion prophylaxis after major abdominal surgery by specific observation of two major complications of abdominal surgery (wound healing impairment, and/or postoperative peritonitis) in comparison to a control group.

Secondary Objectives:

* To further evaluate the safety of A-Part® Gel by comparing the incidences of adverse events between the treatment groups (with special attention to anastomosis leakage)
* To explore the efficacy of A-Part® Gel in reducing post-surgical adhesions after median laparotomy

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, who are candidates for a primary and elective median abdominal incision with a length of ≥ 15 cm 2.
* Age ≥ 18 years
* Patients who are legally capable and able to understand the nature, significance and consequences of the study and are willing and able to comply with the study protocol and the follow up
* Written informed consent obtained according to international guidelines and local law. Informed consent will be documented by the volunteer's dated signature, which will be also signed and dated by the investigator
* Patients with an expected survival time >12 months
* For female adults of reproductive potential: Negative pregnancy test at visit 1 and sufficient contraception from time of written consent up to at least 4 months

Exclusion Criteria:

* Patients with a previous median laparotomy and any other abdominal surgery (exceptions: previous laparoscopic appendectomy, cholecystectomy, inguinal hernia repair, gynecological tube sterilisation)
* Patients with a known history of adhesions or a known history of peritonitis
* Patients with a known sensitivity to polyvinylalcohol and/or carboxymethylcellulose
* Simultaneous participation of the patient in another clinical trial or participation in a clinical trial within the last 30 days prior to signing the Informed consent form
* Patients with ASA > 3 or emergency patients (including severe psychic diesease)
* Patients with ascites > 200 ml
* Patients with peritoneal carcinosis or peritoneal dialysis
* Patients with a diagnosed peritonitis, intra-abdominal abscess or other intra-abdominal infection
* Patient with renal impairment (Creatinine > 1.3 mg/dl)
* Patients with systemic immunosuppression (e.g. hydrocortisone > 50mg daily [oral/i.v.] at any day or any equivalent dosage; other immunosuppressants like Azathioprin, Mycophenolatmofetil, Ciclosporin, Everolimus, Methotrexat, ect.), chemotherapy or radiotherapy within the last 2 weeks prior to surgery
* Surgical procedures or patient characteristics which require insertion of more than 2 intra-abdominal drainages
* Women within a pregnancy or breast-feeding mothers or women who wish to get pregnant within the next 4 months after surgery or women without sufficient contraceptive care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-07; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of wound healing impairment and/or postoperative peritonitis after surgery | 28 (+10) days

SECONDARY OUTCOMES:
Occurrence of anastomosis leakage after surgery | within 28 (+10) days
Occurrence of adverse events (AEs) and serious adverse events (SAEs) after surgery | postoperative hospital stay and up to 3 months
Adhesion rates along the scar examined by ultrasound-assessment | 14 days (range: day 7-14), 28 days (+10 days), 3 months (± 14 days)

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Walter Jauch, Prof.Dr., Principal Investigator — Chirurgische Klinik und Poliklinik - Großhadern, Klinikum der Universität München
Locations (1):
- Chirurgische Klinik und Poliklinik - Großhadern, Klinikum der Universitaet Muenchen, Munich, Bavaria, Germany

REFERENCES:
- [Background] Ellis H. Wound repair. Reaction of the peritoneum to injury. Ann R Coll Surg Engl. 1978 May;60(3):219-21. No abstract available. PMID 646316
- [Background] Parker MC, Ellis H, Moran BJ, Thompson JN, Wilson MS, Menzies D, McGuire A, Lower AM, Hawthorn RJ, O'Briena F, Buchan S, Crowe AM. Postoperative adhesions: ten-year follow-up of 12,584 patients undergoing lower abdominal surgery. Dis Colon Rectum. 2001 Jun;44(6):822-29; discussion 829-30. doi: 10.1007/BF02234701. PMID 11391142
- [Background] Ellis H. Intraabdominal and postoperative peritoneal adhesions. J Am Coll Surg. 2005 May;200(5):641-4. doi: 10.1016/j.jamcollsurg.2004.10.023. No abstract available. PMID 15848353
- [Background] Parker MC, Wilson MS, Menzies D, Sunderland G, Clark DN, Knight AD, Crowe AM; Surgical and Clinical Adhesions Research (SCAR) Group. The SCAR-3 study: 5-year adhesion-related readmission risk following lower abdominal surgical procedures. Colorectal Dis. 2005 Nov;7(6):551-8. doi: 10.1111/j.1463-1318.2005.00857.x. PMID 16232234
- [Background] Gomel V. Reproductive surgery. Minerva Ginecol. 2005 Feb;57(1):21-8. PMID 15758863
- [Background] Fazio VW, Cohen Z, Fleshman JW, van Goor H, Bauer JJ, Wolff BG, Corman M, Beart RW Jr, Wexner SD, Becker JM, Monson JR, Kaufman HS, Beck DE, Bailey HR, Ludwig KA, Stamos MJ, Darzi A, Bleday R, Dorazio R, Madoff RD, Smith LE, Gearhart S, Lillemoe K, Gohl J. Reduction in adhesive small-bowel obstruction by Seprafilm adhesion barrier after intestinal resection. Dis Colon Rectum. 2006 Jan;49(1):1-11. doi: 10.1007/s10350-005-0268-5. PMID 16320005
- [Background] Yamaoka T, Takahashi Y, Fujisato T, Lee CW, Tsuji T, Ohta T, Murakami A, Kimura Y. Novel adhesion prevention membrane based on a bioresorbable copoly(ester-ether) comprised of poly-L-lactide and Pluronic: in vitro and in vivo evaluations. J Biomed Mater Res. 2001 Mar 15;54(4):470-9. doi: 10.1002/1097-4636(20010315)54:43.0.co;2-x. PMID 11426591
- [Background] Diamond MP, Freeman ML. Clinical implications of postsurgical adhesions. Hum Reprod Update. 2001 Nov-Dec;7(6):567-76. doi: 10.1093/humupd/7.6.567. PMID 11727865
- [Background] Becker JM, Stucchi AF. Intra-abdominal adhesion prevention: are we getting any closer? Ann Surg. 2004 Aug;240(2):202-4. doi: 10.1097/01.sla.0000133118.38686.d0. No abstract available. PMID 15273541
- [Background] Treutner KH, Bertram P, Loser S, Winkeltau G, Schumpelick V. [Prevention and therapy of intra-abdominal adhesions. A survey of 1,200 clinics in Germany]. Chirurg. 1995 Apr;66(4):398-403. German. PMID 7634953
- [Background] Holmdahl L, Risberg B, Beck DE, Burns JW, Chegini N, diZerega GS, Ellis H. Adhesions: pathogenesis and prevention-panel discussion and summary. Eur J Surg Suppl. 1997;(577):56-62. PMID 9076453
- [Background] Sjosten AC, Blomgren H, Larsson B, Edelstam GA. Precautions taken to prevent adhesions--a questionnaire study among Swedish obstetricians and gynaecologists. Eur J Surg. 1999 Aug;165(8):736-41. doi: 10.1080/11024159950189492. PMID 10494637
- [Background] Trickett JP, Rainsbury RM, Green R. Paradoxical outcome after use of hyaluronate barrier to prevent intra-abdominal adhesions. J R Soc Med. 2001 Apr;94(4):183-4. doi: 10.1177/014107680109400408. No abstract available. PMID 11317621
- [Background] Besheer A, Mader K, Kaiser S, Kressler J, Weis C, Odermatt EK. Tracking the urinary excretion of high molar mass poly(vinyl alcohol). J Biomed Mater Res B Appl Biomater. 2007 Aug;82(2):383-9. doi: 10.1002/jbm.b.30743. PMID 17238166
- [Background] Kaneo Y, Hashihama S, Kakinoki A, Tanaka T, Nakano T, Ikeda Y. Pharmacokinetics and biodisposition of poly(vinyl alcohol) in rats and mice. Drug Metab Pharmacokinet. 2005 Dec;20(6):435-42. doi: 10.2133/dmpk.20.435. PMID 16415529
- [Background] Yamaoka T, Tabata Y, Ikada Y. Fate of water-soluble polymers administered via different routes. J Pharm Sci. 1995 Mar;84(3):349-54. doi: 10.1002/jps.2600840316. PMID 7616376
- [Background] Yamaoka T, Tabata Y, Ikada Y. Comparison of body distribution of poly(vinyl alcohol) with other water-soluble polymers after intravenous administration. J Pharm Pharmacol. 1995 Jun;47(6):479-86. doi: 10.1111/j.2042-7158.1995.tb05835.x. PMID 7674130
- [Background] Ito T, Yeo Y, Highley CB, Bellas E, Benitez CA, Kohane DS. The prevention of peritoneal adhesions by in situ cross-linking hydrogels of hyaluronic acid and cellulose derivatives. Biomaterials. 2007 Feb;28(6):975-83. doi: 10.1016/j.biomaterials.2006.10.021. Epub 2006 Nov 15. PMID 17109954
- [Background] Beck DE, Cohen Z, Fleshman JW, Kaufman HS, van Goor H, Wolff BG; Adhesion Study Group Steering Committee. A prospective, randomized, multicenter, controlled study of the safety of Seprafilm adhesion barrier in abdominopelvic surgery of the intestine. Dis Colon Rectum. 2003 Oct;46(10):1310-9. doi: 10.1007/s10350-004-6739-2. PMID 14530667
- [Background] Salum M, Wexner SD, Nogueras JJ, Weiss E, Koruda M, Behrens K, Cohen S, Binderow S, Cohen J, Thorson A, Ternent C, Christenson M, Blatchford G, Pricolo V, Whitehead M, Doveney K, Reilly J, Glennon E, Larach S, Williamson P, Gallagher J, Ferrara A, Harford F, Fry R, Eisenstat T, Notaro J, Chinn B, Yee L, Stamos M, Cole P, Dunn G, Singh A; Program Directors Association in Colon and Rectal Surgery. Does sodium hyaluronate- and carboxymethylcellulose-based bioresorbable membrane (Seprafilm) decrease operative time for loop ileostomy closure? Tech Coloproctol. 2006 Oct;10(3):187-90; discussion 190-1. doi: 10.1007/s10151-006-0278-x. Epub 2006 Sep 20. PMID 16969618
- [Background] Kusunoki M, Ikeuchi H, Yanagi H, Noda M, Tonouchi H, Mohri Y, Uchida K, Inoue Y, Kobayashi M, Miki C, Yamamura T. Bioresorbable hyaluronate-carboxymethylcellulose membrane (Seprafilm) in surgery for rectal carcinoma: a prospective randomized clinical trial. Surg Today. 2005;35(11):940-5. doi: 10.1007/s00595-005-3061-0. PMID 16249848
- [Background] Weis C, Odermatt EK, Kressler J, Funke Z, Wehner T, Freytag D. Poly(vinyl alcohol) membranes for adhesion prevention. J Biomed Mater Res B Appl Biomater. 2004 Aug 15;70(2):191-202. doi: 10.1002/jbm.b.30007. PMID 15264300
- [Background] McLeod R. Does Seprafilm really reduce adhesive small bowel obstructions? Dis Colon Rectum. 2006 Aug;49(8):1234; author reply 1235-6. doi: 10.1007/s10350-006-0621-3. No abstract available. PMID 16826328
- [Background] Hyman NH. Justifiable conclusions? Dis Colon Rectum. 2006 Aug;49(8):1236-7; author reply 1237-8. doi: 10.1007/s10350-006-0623-1. No abstract available. PMID 16845562
- [Background] Hadaegh A, Burns J, Burgess L, Rose R, Rowe E, LaMorte WW, Becker JM. Effects of hyaluronic acid/carboxymethylcellulose gel on bowel anastomoses in the New Zealand white rabbit. J Gastrointest Surg. 1997 Nov-Dec;1(6):569-75. doi: 10.1016/s1091-255x(97)80074-1. PMID 9834393
- [Background] Erturk S, Yuceyar S, Temiz M, Ekci B, Sakoglu N, Balci H, Dirican A, Cengiz A, Saner H. Effects of hyaluronic acid-carboxymethylcellulose antiadhesion barrier on ischemic colonic anastomosis: an experimental study. Dis Colon Rectum. 2003 Apr;46(4):529-34. doi: 10.1007/s10350-004-6594-1. PMID 12682549
- [Background] Schuster C, Wuthrich B, Hartmann K, Kuhn M. Anaphylaxis to E466. Allergy. 2000 Mar;55(3):303-4. doi: 10.1034/j.1398-9995.2000.00401.x. No abstract available. PMID 10753030
- [Background] Arnaud JP, Hennekinne-Mucci S, Pessaux P, Tuech JJ, Aube C. Ultrasound detection of visceral adhesion after intraperitoneal ventral hernia treatment: a comparative study of protected versus unprotected meshes. Hernia. 2003 Jun;7(2):85-8. doi: 10.1007/s10029-003-0116-2. Epub 2003 Feb 25. PMID 12820030
- [Background] Karliczek A, Jesus EC, Matos D, Castro AA, Atallah AN, Wiggers T. Drainage or nondrainage in elective colorectal anastomosis: a systematic review and meta-analysis. Colorectal Dis. 2006 May;8(4):259-65. doi: 10.1111/j.1463-1318.2006.00999.x. PMID 16630227
- [Background] Jesus EC, Karliczek A, Matos D, Castro AA, Atallah AN. Prophylactic anastomotic drainage for colorectal surgery. Cochrane Database Syst Rev. 2004 Oct 18;2004(4):CD002100. doi: 10.1002/14651858.CD002100.pub2. PMID 15495028
- [Background] Menzies D, Pascual MH, Walz MK, Duron JJ, Tonelli F, Crowe A, Knight A; ARIEL Registry. Use of icodextrin 4% solution in the prevention of adhesion formation following general surgery: from the multicentre ARIEL Registry. Ann R Coll Surg Engl. 2006 Jul;88(4):375-82. doi: 10.1308/003588406X114730. PMID 16834859
- [Background] Sorensen LT, Malaki A, Wille-Jorgensen P, Kallehave F, Kjaergaard J, Hemmingsen U, Moller LN, Jorgensen T. Risk factors for mortality and postoperative complications after gastrointestinal surgery. J Gastrointest Surg. 2007 Jul;11(7):903-10. doi: 10.1007/s11605-007-0165-4. PMID 17468915
- [Background] Guenaga KF, Matos D, Castro AA, Atallah AN, Wille-Jorgensen P. Mechanical bowel preparation for elective colorectal surgery. Cochrane Database Syst Rev. 2005 Jan 25;(1):CD001544. doi: 10.1002/14651858.CD001544.pub2. PMID 15674882
- [Background] Blackwelder WC. "Proving the null hypothesis" in clinical trials. Control Clin Trials. 1982 Dec;3(4):345-53. doi: 10.1016/0197-2456(82)90024-1. PMID 7160191
- [Background] Lang R, Baumann P, Jauch KW, Schmoor C, Weis C, Odermatt E, Knaebel HP. A prospective, randomised, controlled, double-blind phase I-II clinical trial on the safety of A-Part Gel as adhesion prophylaxis after major abdominal surgery versus non-treated group. BMC Surg. 2010 Jul 6;10:20. doi: 10.1186/1471-2482-10-20. PMID 20604918
- [Result] Lang R, Baumann P, Schmoor C, Odermatt EK, Wente MN, Jauch KW. A-Part Gel, an adhesion prophylaxis for abdominal surgery: a randomized controlled phase I-II safety study [NCT00646412]. Ann Surg Innov Res. 2015 Sep 2;9:5. doi: 10.1186/s13022-015-0014-1. eCollection 2015. PMID 26336510